CLINICAL TRIAL: NCT05732389
Title: Immunotherapy in Patients With Early dMMR Rectal Cancer
Acronym: RESET-R
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: Rigshospitalet, Denmark (Other); Zealand University Hospital (Other); Aalborg University Hospital (Other); Aarhus University Hospital (Other); Bispebjerg Hospital (Other); Herlev and Gentofte Hospital (Other); Vejle Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KFE nr. 22.20
Record Dates: First submitted 2023-01-17; First posted 2023-02-17 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Cancer of Rectum
MeSH Terms: conditions — Rectal Neoplasms | interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- nivolumab + ipilimumab (Experimental): Patients will be treated with 1 or 2 cycles of combination immunotherapy:
  Cycle 1: Nivolumab 3 mg/kg days 1 and 15 & ipilimumab 1 mg/kg day 1 Cycle 2: Nivolumab 3 mg/kg days 50 and 65 & ipilimumab 1 mg/kg day 50
  Interventions: Drug: Nivolumab; Drug: Ipilimumab

INTERVENTIONS:
Drug: Nivolumab — Nivolumab is a highly selective fully humanized, IgG4 monoclonal antibody inhibitor of programmed death-1 (PD-1) (17). PD-1 is an inhibitory receptor expressed on the surface of T-cells, B cells, macrophages, and NK cells. Endogenous binding of PD-1 with one of its two ligands PD-L1 and PD-L2 results in production of an inhibitory signal which results in reduction of T-cell proliferation, cytokine production, and cytotoxic activity. This results in significant dampening of the immune response. Nivolumab acts to selectively block the receptor activation of PD-L1 and PD-L2, resulting in a release of PD-1 mediated inhibition of the immune response.
  Other Names: Opdivo
Drug: Ipilimumab — Ipilimumab is a fully humanized monoclonal anti-CTLA-4 antibody that acts as an antineoplastic ICI by selectively binding to cytotoxic T-lymphocyte-associated antigen 4, a molecule located on the surface of cytotoxic T-cells, suppressing the immune response (17). Ipilimumab blocks CTLA-4, leading to a continuously active immune response in malignant cells.
  Other Names: Yervoy

SUMMARY:
The purpose of this investigator-initiated, multicenter phase II trial is to evaluate the efficacy and tolerability of nivolumab and ipilimumab in patients with stage 1-3 MSI/dMMR rectal cancer.

The primary objective is:

Number of patients with complete clinical response after one or two cycles of immunotherapy.

Patients will be treated with 1 or 2 cycles of combination immunotherapy:

Cycle 1: Nivolumab 3 mg/kg days 1 and 15 & ipilimumab 1 mg/kg day 1 Cycle 2: Nivolumab 3 mg/kg days 50 and 65 & ipilimumab 1 mg/kg day 50

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Histologically verified non-metastatic rectal cancer stage 1-3.
* No indication for local therapy like TEM.
* Histologically verified dMMR or MSI.
* Performance status (WHO) of 0-1.
* No previous chemotherapy, radiotherapy or immunotherapy for colorectal cancer
* Adequate haematological function defined as neutrophils ≥ 1.5 x 109/l and platelets ≥ 100 x 109/l.
* Adequate organ function (bilirubin ≤ 1.5 x UNL (upper normal limit), GFR (may be calculated) > 30 ml/min.
* Women of childbearing potential must have been tested negative in a serum pregnancy test within five days prior to registration. Fertile patients must agree to use a highly effective method of birth control. (i.e., pregnancy rate of less than 1 % per year) (Appendix 1) during the study and for six months after the discontinuation of study medication.
* Has provided written informed consent prior to performance of any study procedure.
* Written informed consent must be obtained according to the local Ethics Committee requirements.

Exclusion Criteria:

* Any other condition or therapy, which in the investigator's opinion may pose a risk to the patient or interfere with the study objectives.
* Concomitant use of systemic glucocorticoids more than the equivalent dose to tablet prednisolone 10 mg/day. Treatment with systemic glucocorticoids must end no later than two weeks before inclusion.
* Subjects with active, known, or suspected autoimmune disease. Subjects with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enrol.
* Known allergy or intolerance to any of the drugs used (nivolumab and ipilimumab).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2052-02 (Estimated)

PRIMARY OUTCOMES:
Complete clinical response | Evaluated at day 93 (+/- 7 days) after one or two cycles of immunotherapy. (Each cycle is 7 weeks)
  Proportion of patients with complete clinical response Complete clinical response will be defined as no visible or palpable tumor examined by rectal exploration (if low tumors), endoscopy and MR-scan. Patients with definite but less than complete regression BUT with a representative biopsy without viable tumor cells will also be classified as cCR in this trial.

SECONDARY OUTCOMES:
Complete biological response | Evaluated at day 93 (+/- 7 days) after one or two cycles of immunotherapy. (Each cycle is 7 weeks)
  Proportion of patients with complete biological response
12 months recurrence | after 12 months
  Proportion of patients without any sign of recurrence after 12 months.
Respons rate | after 1 or 2 cycles of immunotherapy. (Each cycle is 7 weeks)
  Response rate according to mrTRG.
Adverse events | after 1 or 2 cycles of immunotherapy and months 4, 10, 16, and 24. (Each cycle is 7 weeks)
  Adverse events assessed by the investigator according to the definitions in NCI-CTC, version 5.0
Bio-marker predictive models for treatment response and survival. | after 1 or 2 cycles of immunotherapy. (Each cycle is 7 weeks)
  Correlation between bio-markers (ctDNA and CEA) and outcome.
Quality of life (EORCT QLQ-C30) | after 1 or 2 cycles of immunotherapy and months 4, 10, 16, and 24. (Each cycle is 7 weeks)
  Change in Quality of life (EORCT QLQ-C30)
Quality of life (EORCT QLQ-CR29) | after 1 or 2 cycles of immunotherapy and months 4, 10, 16, and 24. (Each cycle is 7 weeks)
  Change in Quality of life (EORCT QLQ-CR29)

CONTACTS AND LOCATIONS:
Overall Officials: Line S Tarpgaard, MD, Phd, Principal Investigator — Department of Oncology, Odense University Hospital, Denmark
Locations (5):
- Denmark (5):
  - Aalborg University Hospital, Aalborg
  - Aarhus University Hospital, Aarhus
  - Rigshospitalet, Copenhagen
  - Department of Oncology, Odense University Hospital, Odense
  - Zealand University Hospital, Roskilde

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol (2022-10-30): https://cdn.clinicaltrials.gov/large-docs/89/NCT05732389/Prot_000.pdf